CLINICAL TRIAL: NCT02381925
Title: Multicenter Registry Comparing Preoperative Imaging for Primary Hyperparathyroidism
Status: Withdrawn | Type: Observational
Why Stopped: The study never opened due to funding issues
Sponsor: Duke University (Other)
Collaborators: University of California, Los Angeles (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00061739
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Parathyroid Adenoma
Keywords: CT; Scintigraphy; Ultrasound
MeSH Terms: conditions — Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims are:

1. To compare the diagnostic performance of parathyroid four-dimensional CT (4D-CT), scintigraphy, and ultrasound in patients who underwent parathyroid surgery for primary hyperparathyroidism.
2. To compare 4D-CT, scintigraphy, and ultrasound for the ability to perform focused parathyroidectomy, and for rates of persistent hyperparathyroidism and complications from parathyroid surgery.

Methods The investigators will create a multicenter registry consisting of patients having parathyroid surgery for primary hyperparathyroidism from July 2009 to June 2016. Initial participating centers include Duke University Medical Center, University California Los Angeles (UCLA) and University of Arkansas for Medical Sciences (UAMS).

There will be no intervention in the patient's treatment or imaging. The management will be determined by the surgeon or clinician supervising the patient's care.

The registry will consist of patient data regarding basic demographics, history of prior neck/chest surgery or radiation, parathyroid imaging, biochemical evaluation, intraoperative surgical findings, parathyroid pathology, and surgical outcomes within the first 6 months (persistent disease, recurrent laryngeal nerve injury, and hypoparathyroidism). Data will be entered into REDCap with no PHI. The investigators expect to include 3000 patients in the registry (1000 from Duke).

ELIGIBILITY:
Inclusion Criteria:

* patients having parathyroid surgery for primary hyperparathyroidism from July 2009 to June 2016

Exclusion Criteria:

* age less than 18 years
* parathyroid carcinoma
* secondary or tertiary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will include all patients, aged 18 years or older, who underwent parathyroid surgery from July 2009 to July 2016.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance of imaging | 6 months

SECONDARY OUTCOMES:
ability to perform focused parathyroidectomy | 6 months
rates of persistent hyperparathyroidism after parathyroidectomy | 6 months
parathyroidectomy surgical complications | 6 months